CLINICAL TRIAL: NCT05722626
Title: The Effects of Intra-articular Platelet-Rich Plasma Injection on The Severity of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Bali Internasional (Other)
Responsible Party: Principal Investigator, Ida Ayu Ratih Wulansari Manuaba, Ida Ayu Ratih Wulansari Manuaba, Universitas Bali Internasional
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01_028/UNBI/EC/V/2021
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet-rich plasma (Experimental): PRP manufactured by T_Biyoteknoloji LTD, Turkey
  Interventions: Procedure: PRP
- Normal Saline (Placebo Comparator): NaCl 0.9%
  Interventions: Other: Normal Saline

INTERVENTIONS:
Procedure: PRP — 2 ml of platelet rich plasma intraarticular injection twice in one week interval
  Other Names: T_Biyoteknoloji LTD, Turkey
  Arms: Platelet-rich plasma
Other: Normal Saline — NaCl 0.9%
  Other Names: NaCl 0.9%
  Arms: Normal Saline

SUMMARY:
This is a single-center, randomized control trial The aim of this study is to compare PRP with placebo as the treatment of knee OA Conducted at Puri Raharja Hospital Bali in January-June 2022 Sample consisted of 106 patients with knee OA grades 2-3 Kellgren-Lawrence, randomized into PRP group and placebo group Samples were injected with 2 ml PRP or normal saline twice at one-week interval The severity of knee OA was assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) before injection and two weeks after the first injection.

ELIGIBILITY:
Inclusion Criteria:

patients with knee pain for at least three months, aged between 40 to 80 years old, and whose results of radiological examination of the knee indicated OA grades 2-4 based on the Kellgren Lawrence classification

Exclusion Criteria:

polyarticular rheumatic disease; knee arthroscopy <1 year; intra-articular injection of hyaluronic acid (HA) or steroids in the past three months; current infection, diabetes, rheumatoid arthritis, coagulopathy disorders, anticoagulant or antiplatelet aggregation therapy, immunodeficiency disease, taking non-steroidal anti-inflammatory drugs (NSAIDs) two weeks prior to the procedure, knee trauma; inflammation; and tumors around the knee

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
WOMAC | 2 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) based on questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anak Agung Sagung Mirah Prabandari, dr., Principal Investigator — Warmadewa University
Locations (1):
- Puri Raharja Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No